CLINICAL TRIAL: NCT04873362
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Efficacy and Safety of Adjuvant Atezolizumab or Placebo and Trastuzumab Emtansine for HER2-Positive Breast Cancer at High Risk of Recurrence Following Preoperative Therapy
Brief Title: A Study Evaluating the Efficacy and Safety of Adjuvant Atezolizumab or Placebo and Trastuzumab Emtansine for Participants With HER2-Positive Breast Cancer at High Risk of Recurrence Following Preoperative Therapy
Acronym: Astefania
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WO42633; 2020-003681-40 (EudraCT Number); 2023-503568-18-00 (EU CTIS Number)
Record Dates: First submitted 2021-04-21; First posted 2021-05-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — atezolizumab; Ado-Trastuzumab Emtansine; Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Placebo + Trastuzumab Emtansine (Active Comparator): Participants will receive an intravenous (IV) infusion of placebo prior to the IV infusion of trastuzumab emtansine on Day 1 of each 21-day cycle for a total of 14 cycles.
  Interventions: Drug: Trastuzumab Emtansine; Drug: Placebo; Drug: Trastuzumab
- Arm B: Atezolizumab + Trastuzumab Emtansine (Experimental): Participants will receive an IV infusion of atezolizumab prior to the IV infusion of trastuzumab emtansine on Day 1 of each 21-day cycle for a total of 14 cycles.
  Interventions: Drug: Atezolizumab; Drug: Trastuzumab Emtansine; Drug: Trastuzumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a dose of 1200 mg every three weeks (Q3W) for 14 cycles.
  Other Names: Tecentriq, RO5541267, MPDL3280A
  Arms: Arm B: Atezolizumab + Trastuzumab Emtansine
Drug: Trastuzumab Emtansine — Trastuzumab emtansine will be administered at a dose of 3.6 mg/kg Q3W for 14 weeks.
  Other Names: Kadcyla, T-DM1, RO5304020
Drug: Placebo — Placebo matched to atezolizumab will be administered at a dose of 1200 mg Q3W for 14 cycles.
  Arms: Arm A: Placebo + Trastuzumab Emtansine
Drug: Trastuzumab — Trastuzumab will be used to complete 14 cycles of study treatment if trastuzumab emtansine is discontinued for toxicity not considered to be related to the trastuzumab component of the drug.
  Other Names: Herceptin

SUMMARY:
This is a Phase III, two-arm, randomized, double-blind placebo-controlled study in participants with HER2-positive primary breast cancer who have received preoperative chemotherapy and HER2-directed therapy, including trastuzumab followed by surgery, with a finding of residual invasive disease in the breast and/or axillary lymph nodes.

As of June 4, 2024, this study is no longer accepting any newly screened participants.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast carcinoma
* Centrally-confirmed human epidermal growth factor receptor 2 (HER2)-positive invasive breast cancer
* Centrally confirmed PD-L1 and hormone receptor status
* Clinical stage at disease presentation (prior to neoadjuvant therapy): cT4/anyN/M0, any cT/N2-3/M0, or cT1-3/N0-1/M0 (participants with cT1mi/T1a/T1b/N0 are not eligible)
* Completion of pre-operative systemic chemotherapy including at least 9 weeks of taxane and 9 weeks of trastuzumab (anthracycline and/or additional HER2-targeted agents are permitted)
* <=12 weeks between primary surgery and randomization
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Screening left ventricular ejection fraction (LVEF) >= 50% and no decrease in LVEF by >15% from the pre-chemotherapy LVEF. If no pre-chemotherapy LVEF, screening LVEF >= 55%
* Life expectancy >= 6 months
* Adequate hematologic and end organ function

Exclusion Criteria:

* Stage IV breast cancer
* An overall response of disease progression according to the investigator at the conclusion of preoperative systemic therapy
* Prior treatment with T-DM1, or atezolizumab, or other immune checkpoint inhibitors
* History of exposure to various cumulative doses of anthracyclines
* History of other malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or ductal carcinoma in situ (DCIS)
* Current grade >=2 peripheral neuropathy
* History of idiopathic pulmonary fibrosis, organizing pneumonia, or pneumonitis
* History of or active autoimmune disease or immune deficiency
* Treatment with immunostimulatory or immunosuppressive agents
* Cardiopulmonary dysfunction
* Any known active liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1188 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2034-10-02 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-free Survival (IDFS) in the Full Analysis Set (FAS) | From baseline until the first occurrence of iDFS event or death, through primary analysis data cut off (approximately 7 years)
  IDFS event is defined as the time from randomization to the first occurrence of the following events: ipsilateral invasive breast tumor recurrence, ipsilateral local-regional invasive breast cancer recurrence, contralateral invasive breast cancer, distant recurrence, death from any cause.

SECONDARY OUTCOMES:
IDFS Including Second Primary Non-breast Invasive Cancer | From baseline until the first occurrence of iDFS event or death, through the end of study (approximately 10 years from last participant in [LPI])
IDFS in the PD-L1-positive and the PD-L1-negative Population | From baseline until the first occurrence of iDFS event or death, through the end of study (approximately 10 years from LPI)
  Defined as all randomized participants from the ITT population with a centrally assessed PD-L1-positive [i.e., PD-L1 status of IC1/2/3] or PD-L1-negative status [i.e.,PD-L1 status of IC0] at randomization as per corresponding stratification factors recorded in the interactive web-based response system (IWRS).
Disease-free Survival (DFS) | From baseline until the first occurrence of DFS event or death, through the end of study (approximately 10 years from LPI)
Overall Survival (OS) | From baseline to death from any cause through the end of study (approximately 10 years from LPI)
Distant Recurrence-free Interval (DRFI) | From baseline until distant disease recurrence, through the end of study (approximately 10 years from LPI)
Number of Participants with Clinically Meaningful Deterioration in Global Health Status/Quality of Life (GHS/QoL) Physical, Role, and Cognitive Function | From baseline until 2 years after study treatment completion/discontinuation visit (approximately 3 years)
  Clinically Meaningful Deterioration will be Measured by Scales of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer (EORTC QLQ C30)
Mean Absolute Scores in GHS/QoL, Physical, Role, and Cognitive Function, as Assessed Using the EORTC QLQ-C30 | From baseline until 2 years after study treatment completion/discontinuation visit (approximately 3 years)
  The European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 Questionnaire (EORTC QLQ-C30) is a self-reported measure. Functioning and symptoms items are scored on a 4-point scale: 1=Not at all, 2=A little, 3=Quite a bit, 4=Very much. GHS and QoL items are scored on a 7-point scale: 1=Very poor, 2, 3, 4, 5, 6, 7=Excellent. Scores will be transformed to a range of 0 to 100, with higher scores (i.e. closer to 100) reflecting better functioning, better GHS/QoL, and worse symptoms.
Mean Change From Baseline Scores in GHS/QoL, Physical, Role, and Cognitive Function, as Assessed Using the EORTC QLQ-C30 | From baseline until 2 years after study treatment completion/discontinuation visit (approximately 3 years)
  The European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 Questionnaire (EORTC QLQ-C30) is a self-reported measure. Functioning and symptoms items are scored on a 4-point scale: 1=Not at all, 2=A little, 3=Quite a bit, 4=Very much. GHS and QoL items are scored on a 7-point scale: 1=Very poor, 2, 3, 4, 5, 6, 7=Excellent. Scores will be transformed to a range of 0 to 100, with higher scores (i.e. closer to 100) reflecting better functioning, better GHS/QoL, and worse symptoms.
Percentage of Participants with Adverse Events (AEs) According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0) | From baseline up to 10 years
Maximum Serum Concentrations (Cmax) for Atezolizumab | Day 1 of Cycles 1 and 4 after 30 minutes post-infusion (a cycle=21 days)
Minimum Serum Concentrations (Cmin) for Atezolizumab | Pre-infusion on Day 1 of Cycles 1, 2, 3, 4 and 8 (a cycle=21 days) and at study treatment completion/discontinuation visit (approximately 11 months after Cycle 1 Day 1)
Cmax for Trastuzumab Emtansine | Day 1 of Cycles 1 and 4 after 30 minutes post-infusion (a cycle=21 days)
Cmin for Trastuzumab Emtansine | Pre-infusion on Day 1 of Cycles 1 and 4 (a cycle=21 days) and at study treatment completion/discontinuation visit (approximately 11 months after Cycle 1 Day 1)
Cmax for Total Trastuzumab | Day 1 of Cycles 1 and 4 after 30 minutes post-infusion (a cycle=21 days)
Cmin for Total Trastuzumab | Pre-infusion on Day 1 of Cycles 1 and 4 (a cycle=21 days) and at study treatment completion/discontinuation visit (approximately 11 months after Cycle 1 Day 1)
Cmax for DM1 | Day 1 of Cycles 1 and 4 after 30 minutes post-infusion (a cycle=21 days)
  DM1 = a thiol-containing maytansinoid anti-microtubule agent; N2'-deacetyl-N2'-(3-mercapto-1-oxopropyl)-maytansine
Percentage of Participants with Anti-drug Antibodies (ADAs) to Atezolizumab | Pre-infusion on Day 1 of Cycles 1, 2, 3, 4 and 8 (a cycle=21 days) and at study treatment completion/discontinuation visit (approximately 11 months after Cycle 1 Day 1)
Percentage of Participants with ADAs to Trastuzumab Emtansine | Pre-infusion on Day 1 of Cycles 1 and 4 (a cycle=21 days) and at study treatment completion/discontinuation visit (approximately 11 months after Cycle 1 Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (239):
- United States (22):
  - Alabama Oncology, Birmingham, Alabama
  - Roy and Patricia Disney Family Cancer Center- Providence Saint Joseph Medical Center, Buena, California
  - UCLA Medical Center, Santa Monica, California
  - Innovation Clinical Research Institute, Whittier, California
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital, Carrollton, Georgia
  - University of Iowa, Iowa City, Iowa
  - New England Cancer Specialists, Westbrook, Maine
  - The Valley Hospital, Paramus, New Jersey
  - Levine Cancer Institute, Charlotte, North Carolina
  - Abramson Cancer Center; Univ of Pennsylvania; Clinical Research Unit, Philadelphia, Pennsylvania
  - The West Clinic, Germantown, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Mays Cancer Center at UT Health San Antonio MD Anderson Cancer, San Antonio, Texas
  - Hematology Oncology Associates of Fredericksburg, Inc., Fredericksburg, Virginia
  - Virginia Oncology Associates - New Port News, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Oncology Associates - Virginia Beach, Virginia Beach, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Australia (3):
  - Macarthur Cancer Therapy Centre, Campbelltown, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
- Austria (3):
  - Tiroler Landeskrankenanstalten Ges.M.B.H., Innsbruck
  - Ordensklinikum Linz Barmherzige Schwestern, Linz
  - Lkh Salzburg - Univ. Klinikum Salzburg, Salzburg
- Belgium (3):
  - Cliniques Universitaires St-Luc, Brussels
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - Clinique St. Elizabeth, Namur
- Brazil (10):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
  - Núcleo de Pesquisa São Camilo, São Paulo, São Paulo
- Bulgaria (3):
  - COC Plovdiv, Plovdiv
  - Medical Center "Nadezhda Clinical" EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
- China (13):
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital - Sichuan University, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - Sun Yat-sen Memorial Hospital, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affilicated Hospital, Sun Yat-sen University, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Zhongshan Hospital Fudan University, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - Zhejiang Cancer Hospital, Zhejiang
  - Henan Cancer Hospital, Zhengzhou
- Czechia (6):
  - Masaryk?v onkologický ústav, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Nemocnice AGEL Novy Jicin a.s., Nový Jičín
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni Poliklinika Vseobecne Fakultni Niemocnice, Prague
  - Fakultni Thomayerova nemocnice, Praha 4 - Krc
- Vejle Sygehus, Vejle, Denmark
- France (12):
  - Institut Sainte Catherine, Avignon
  - CHRU Besançon, Besançon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CHU Brest Hopital La Cavale Blanche, Brest
  - Centre Francois Baclesse, Caen
  - Groupe Hospitalier Public Du Sud De L'Oise GHPSO, Creil
  - CLCC Leon Berard Lyon, Lyon
  - Centre Hospitalier Uni Ire Caremeau, Nîmes
  - Groupe Hospitalier Diaconesses, Paris
  - Institut Curie, Paris
  - Pole Regional De Cancerologie, Poitiers
  - HOPITAL RENE HUGUENIN, Institut Curie, Saint-Cloud
- Germany (19):
  - Klinikum Augsburg, Augsburg
  - Hochwaldkrankenhaus, Bad Nauheim
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Gynäkologisches Zentrum Bonn, Bonn
  - Marienhospital Bottrop, Bottrop
  - Städtisches Klinikum Dessau, Dessau
  - Gynonco Düsseldorf, MVZ Medical Center GmbH, Düsseldorf
  - Frauenarztpraxis Dr. Apel, Dr. Kolpin, Erfurt
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH, Essen
  - AGAPLESION Markus-Krankenhaus, Frankfurt
  - Klinik Johann Wolfgang von Goethe Uni, Frankfurt
  - Praxis für Interdisziplinäre Onkologie und Hämatologie GbR, Freiburg im Breisgau
  - Diakovere Henriettenstift, Frauenklinik, Hanover
  - UNI-Klinikum Campus Kiel Klinik für Gynäkologie und Geburtshilfe, Kiel
  - Städtische Klinik Lüneburg, Lüneburg
  - Klinik & Poliklinik für Frauenheilkunde und Geburtshilfe, Campus Innenstadt, München
  - Klinikum Ernst von Bergmann, Potsdam
  - Leopoldina Krankenhaus der Stadt Schweinfurt GmbH, Schweinfurt
  - Gemeinschaftspraxis für Hämatologie und Onkologie Dr. Reichert/Dr.Janssen, Westerstede
- Greece (6):
  - Anticancer Hospital Ag. Savas, Athens
  - Alexandras General Hospital of Athens, Athens
  - University General Hospital of Heraklion, Crete
  - University Hospital of Larissa, Larissa
  - Metropolitan Hospital, Piraeus
  - European Interbalkan Medical Center, Thessaloniki
- Hong Kong (3):
  - Queen Mary Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- Hungary (3):
  - Budapesti Szent Margit Korhaz, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- India (9):
  - Hemato Oncology Clinic Ahmedabad Pvt Ltd, Ahmedabad, Gujarat
  - Manipal Hospital, Bangalore, Karnataka
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Sahyadri Super Specialty Hospital Hadapsar, Pune, Maharashtra
  - Rajiv Gandhi Cancer Institute & Research Center, New Delhi, National Capital Territory of Delhi
  - Max Super Speciality Hospital, North WEST Delhi, National Capital Territory of Delhi
  - Christian Med Clg & Hspt, Ratnagiri Kilminnal, Tamil Nadu
  - TATA Medical Centre, Kolkata, West Bengal
- Italy (11):
  - AORN'S.G.Moscati, Avellino, Campania
  - U.O.C. Oncologia Medica Senologica, Napoli, Campania
  - Università degli Studi Federico II, Napoli, Campania
  - A.O. Universitaria Policlinico Di Modena, Modena, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO), Aviano, Friuli Venezia Giulia
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Asst Degli Spedali Civili Di Brescia, Brescia, Lombardy
  - Ospedale San Raffaele, Milan, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Ospedale Civile - Livorno, Livorno, Tuscany
  - Azlenda Ospendaliero-Universitaria Pisana, Pisa, Tuscany
- The Aga Khan University-Kenya., Nairobi, Kenya
- Mexico (6):
  - Investigacion Oncofarmaceutica, La Paz, Baja California Sur
  - Instituto Nacional De Cancerologia, Distrito Federal, Mexico CITY (federal District)
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - Centro Medico Dalinde, Mexico City, Mexico CITY (federal District)
  - Filios Alta Medicina, Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City, Oaxaca
- Auckland City Hospital, Cancer and Blood Research, Auckland, New Zealand
- Poland (6):
  - Bialostockie Centrum Onkologii, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Narodowy Instytut Onkologii Odzia? w Gliwicach, Gliwice
  - Szpital Uniwersytecki w Krakowie, Oddzia? Kliniczny Kliniki Onkologii, Krakow
  - Wielkopolskie Centrum Onkologii, Poznan
  - Centrum Onkologii Instytut im.M. Sklodowskiej-Curie, Warsaw
- Portugal (4):
  - Hospital CUF Tejo, Lisbon
  - Hospital de Santa Maria, Lisbon
  - Hospital Beatriz Angelo, Loures
  - IPO do Porto, Porto
- Romania (6):
  - Filantropia Clinical Hospital, Bucharest
  - Amethyst Cluj, Cluj County
  - Cluj-Napoca Emergency Clinical County Hospital, Cluj-Napoca
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Centrul de Oncologie Sfantul Nectarie, Craiova
  - Oncomed SRL, Timișoara
- Russia (13):
  - FSBI Russian Oncology Research Center n.a. Blokhin of MOH RF, Moscow, Moscow Oblast
  - MEDSI Clinical Hospital on Pyatnitsky Highway, Moscow, Moscow Oblast
  - SBIH "Moscow Clinical Scientific and Practical Center named after A.S. Loginov of DHM", Moskva, Moscow Oblast
  - Nizhny Novgorod Regional Clinical Oncology Center, Nizhny Novgorod, Niznij Novgorod
  - Republican Clinical Oncological Dispensary of the Ministry of Healthcare, Kazan, Republic of Karelia
  - SBI of Healthcare Leningrad Regional Oncology Dispensary, Saint Peterburg, Sankt-Peterburg
  - Medical Clinic "AB Medical group", Saint Petersburg, Sankt-Peterburg
  - FSBI?National Medical Research Center of Oncology named after N.N.Petrov? MHRF, Saint Petersburg, Sankt-Peterburg
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg, Sankt-Peterburg
  - SBIH Kaluga Region Clinical Oncology Dispensary, Kaluga
  - LLC Medical and Sanitary Unit "Clinician", Novosibirsk
  - Regional Oncology Dispensary, Tomsk
  - Regional Clinical Oncology Hospital, Yaroslavl
- National Cancer Centre, Singapore, Singapore
- South Korea (10):
  - Kyungpook National University Medical Center, Daegu
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (19):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital de Jerez de la Frontera, Jerez de la Frontera, Cadiz
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Juan Ramon Jimenez, Huelva
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico, Jaén
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Quiron de Madrid, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (6):
  - Chia-Yi Christian Hospital, Chiayi City
  - China Medical University Hospital, Taichung
  - National Cheng Kung Uni Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
- Thailand (4):
  - Chulalongkorn Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Srinagarind Hospital, Khon Kaen
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (16):
  - Adana Baskent University Hospital, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Gazi University Medical Faculty, Oncology Hospital, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Antalya Training and Research Hospital, Antalya
  - Ege University Medical Faculty, Bornova, ?zm?r
  - Dicle University Faculty of Medicine, Diyarbakır
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Istanbul Faculty of Medicine, Istanbul
  - Istanbul University Cerrahpasa Faculty of Medicine, Istanbul
  - Medeniyet University Goztepe Training and Research Hospital., Istanbul
  - Katip Celebi University Ataturk Training and Research Hospital, Izmir
  - Inonu University Medical Faculty of Medicine, Malatya
  - Medical Park Seyhan Hospital, Seyhan
  - Ac?badem Altunizade Hastanesi, Üsküdar
- Uganda Cancer Institute, Kampala, Uganda
- Ukraine (6):
  - Uzhgorod Central City Clinical Hospital, Uzhhorod, Katerynoslav Governorate
  - Municipal Noncommercial Institution Regional Center of Oncology, Kharkiv, Kharkiv Governorate
  - Municipal non profit enterprise of Sumy Regional Council Sumy Regional Clinical Oncology Disp, Sumy, Kholm Governorate
  - CI Dnipropetrovsk CMCH #4 of Dnipropetrovsk RC SI Dnipropetrovsk MA of MOHU Ch of Oncology and MR, Dnipropetrovsk
  - Municipal Institution Kirovograd Regional Oncology Dispensary, Kirovograd
  - Kyiv City Clinical Oncological Center, Kyiv
- United Kingdom (12):
  - Blackpool Victoria Hospital, Blackpool
  - Royal Sussex County Hospital, Brighton
  - Addenbrookes Hospital, Cambridge
  - Cheltenham General Hospital, Cheltenham
  - Barts & London School of Med, London
  - University College London Hospital, London
  - Royal Free Hospital, London
  - Royal Marsden Hospital - London, London
  - Christie Hospital NHS Trust, Manchester
  - Mount Vernon Cancer Centre, Northwood
  - Royal Preston Hospital, Preston
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Hurvitz SA, Bachelot T, Bianchini G, Harbeck N, Loi S, Park YH, Prat A, Gilham L, Boulet T, Gochitashvili N, Monturus E, Lambertini C, Nyawira B, Knott A, Restuccia E, Schmid P. ASTEFANIA: adjuvant ado-trastuzumab emtansine and atezolizumab for high-risk, HER2-positive breast cancer. Future Oncol. 2022 Oct;18(32):3563-3572. doi: 10.2217/fon-2022-0485. Epub 2022 Nov 16. PMID 36382554